CLINICAL TRIAL: NCT03383770
Title: Dual Guidance in Regional Anesthesia - Prospective Randomized Study of Needle-nerve Distance in Different Cannulas for Regional Nerve Blockade
Brief Title: Dual Guidance in Regional Anesthesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Jurgen Birnbaum, PD Dr. med.; Consultant Anaesthesiologist, Charite University, Berlin, Germany
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DUAL
Record Dates: First submitted 2017-12-14; First posted 2017-12-26 (Actual); Last update posted 2022-02-04 (Actual); Status verified 2022-01

CONDITIONS: Anesthesia, Local; Anesthesia; Anesthesia; Adverse Effect

STUDY DESIGN:
Intervention Model Description: The selection of the puncture cannula for regional anaesthesia is not up to the performing anaesthetist, as is usual in the clinical standard, but is made randomly on the basis of a random list. The blockade is carried out by two anaesthetists experienced in regional anaesthesia, who have the principle of dual control. The ultrasound image acquired during the blockade is recorded in the form of an ultrasound video for subsequent evaluation. The recorded ultrasound videos are stored pseudonymously on the server of the Klinik für Anästhesiologie m. S. operativ Intensivmedizin reported to the data protection department.
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tuohy (Active Comparator): After a careful disinfection of the puncture site, under sterile conditions and under ultrasonographic control with the application of nerve stimulation (settings: stimulation current primary 2.0 mA with stepwise reduction over 1.0 mA to 0.5 mA, pulse width 0.1 ms, pulse frequency 2 Hz) of the N. ischiadicus blocked by 20 ml ropivacaine 0.75 %. (electrical nerve stimulation and ultrasound) If no motor response can be triggered by stimulation, the closest possible needle-nerve distance is generated at a pulse strength of 1mA and regional anesthesia is performed. (protective nerve stimulation) Subsequently, the transplantation into the supine position and the further procedure specific to the operation (use of other regional procedures in combination or general anaesthesia).
  A tuohy needle is used.
  Interventions: Procedure: Regional Anesthesia Touhy
- Facet (Active Comparator): After a careful disinfection of the puncture site, under sterile conditions and under ultrasonographic control with the application of nerve stimulation (settings: stimulation current primary 2.0 mA with stepwise reduction over 1.0 mA to 0.5 mA, pulse width 0.1 ms, pulse frequency 2 Hz) of the N. ischiadicus blocked by 20 ml ropivacaine 0.75 %. (electrical nerve stimulation and ultrasound) If no motor response can be triggered by stimulation, the closest possible needle-nerve distance is generated at a pulse strength of 1mA and regional anesthesia is performed. (protective nerve stimulation) Subsequently, the transplantation into the supine position and the further procedure specific to the operation (use of other regional procedures in combination or general anaesthesia).
  A facet needle is used.
  Interventions: Procedure: Regional Anesthesia Facet

INTERVENTIONS:
Procedure: Regional Anesthesia Touhy — The patients receive the planned anaesthesia procedure according to the procedure to be performed. Only nerve blockages are carried out, which are considered to be analgesic useful for the planned operations on the basis of typical nerve courses. A touhy cannula is used.
  Arms: Tuohy
Procedure: Regional Anesthesia Facet — The patients receive the planned anaesthesia procedure according to the procedure to be performed. Only nerve blockages are carried out, which are considered to be analgesic useful for the planned operations on the basis of typical nerve courses. A facet cannula is used.
  Arms: Facet

SUMMARY:
Regional anaesthesia is a frequently used procedure. Currently, blockades are increasingly carried out without nerve stimulation. The risk of nerve lesion is about 3 %. Industrial efforts frequently referred to ultrasound optimisation of the regional anaesthesia cannula. In order to optimise patient safety, the benefit of both procedures (stimulation and ultrasound) should be combined and both procedures optimised. In this study, the influence of the needle electrode size on the stimulability of the nerve ischiadicus should be determined.

DETAILED DESCRIPTION:
There are various methods of performing regional anesthesia. In recent years, the focus has been on ultrasound-supported regional anaesthesia, and the stimulation methods that were often used in the past were no longer used or used less frequently. The combination of both methods may be an additional safety aspect and can contribute to an improved blocking quality. In addition to the best possible ultrasound quality, an optimal stimulation quality is also required. The investigators plan to carry out dual-guidance blockages of the ischiadic nerve with various regional anaesthesia needles (manufacturer of the used needles: Pajunk Medical Produkte GmbH, Geisingen, Germany; Teleflex Medical GmbH, Kernen, Germany). All regional anaesthesia cannulae are approved for the planned blockades of humans in Germany.

ELIGIBILITY:
Inclusion Criteria:

* Presence of the written declaration of consent
* Age of at least 18 years
* No participation in another intervention study during participation

Exclusion Criteria:

* present contraindication for the application of regional anesthesia and nerve stimulation
* Cardiac pacemaker/AICD (Automated internal cardioverter defibrillator) carrier
* Known allergies to used medicines
* Patients under 18 years of age
* Ineligible patients
* Missing consent
* Pregnancy/nursing patients
* Classification of patients into class 4 or higher status according to the American Society of Anesthesiologists
* Existing nerve damage in the target area
* Medically treated diabetes mellitus, alcohol abuse or alcohol abuse in the patient's history (using AUDIT)
* Visibility score of the nerve of 3 or more
* Participation in another intervention study during participation
* Accommodation in an institution on the basis of a court or administrative order

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2018-02-05 (Actual); Primary Completion 2019-09-15 (Actual); Study Completion 2019-09-15 (Actual)

PRIMARY OUTCOMES:
Ultrasound distance | duration of blockade, an average of 15 minutes
  Ultrasound-based measurement of needle-nerve distance during the application of the regional anesthesia of the N. ischiadicus during infragluteal access.

SECONDARY OUTCOMES:
Visibility_1 | duration of blockade, an average of 15 minutes
  Ultrasound visibility of needle
Visibility_2 | duration of blockade, an average of 15 minutes
  Ultrasound visibility of nerve
Impedance | duration of blockade, an average of 15 minutes
  Impedance measured by nerve stimulator while progressing the needle
Effect_motor | duration of surgery and recovery unit, an average of 120 minutes
  Effectiveness of the motor blockade measured by possible movement of the foot
Effect_sensoric | duration of surgery and recovery unit, an average of 120 minutes
  Effectiveness of the blockade measured by temperature sensibility testing on the food

OTHER OUTCOMES:
Impedance_Change | duration of blockade, an average of 15 minutes
  Changes in impedance measurement while blockade
Complications | duration of surgery and recovery unit, an average of 120 minutes
  Occurence of complications of regional anesthesia
Contact | duration of blockade, an average of 15 minutes
  Number of Needle-Nerve-Contacts by Ultrasound-measurement

CONTACTS AND LOCATIONS:
Overall Officials: Jürgen Birnbaum, MD, PhD, Principal Investigator — Charite University, Berlin, Germany
Locations (1):
- Charité - Universitätsmedizin Berlin Campus Charité Mitte, Berlin, Deutschland, Germany

IPD SHARING:
Plan to Share IPD: No